CLINICAL TRIAL: NCT05491070
Title: Efficacy Comparison of Different Femoral Vascular Closure Method Following Percutaneous Transcatheter Aortic Valve Implantation
Brief Title: Comparison of Different Vascular Closure Device in TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201711019RINC
Record Dates: First submitted 2018-07-20; First posted 2022-08-08 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-10

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Vascular Closure Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual Proglide (Experimental): Use Two Progilde for closure of femoral artery with large sheath in transfemoral TAVI
  Interventions: Device: Vascular closure device (Angio-Seal, Progilde)
- Progilde + AngioSeal (Experimental): Use Progilde + AngioSeal for closure of femoral artery with large sheath in transfemoral TAVI
  Interventions: Device: Vascular closure device (Angio-Seal, Progilde)

INTERVENTIONS:
Device: Vascular closure device (Angio-Seal, Progilde) — In transfemoral TAVI, vascular closure devices were used for femoral artery wound closure, progilde and angio-seal can be used in wound closure. We aimed to compared the efficacy and safety of different vascular closure device in TAVI

SUMMARY:
Femoral artery approach for transcatheter aortic valve implantation (TAVI) is an ideal approach site. However the closure for femoral artery after transfemoral TAVI is challenging. We aimed to compared the efficacy and safety of Angio-Seal + Proglide vs. Dual Proglide for femoral arteriotomy closure following TAVI

DETAILED DESCRIPTION:
Aortic stenosis (AS) is a common, potentially fatal condition that emerges as a substantial public health burden. The prevalence of AS is as high as 9.8% in those 80 years or older, with an overall prevalence of 2.8% in adults over 75 years of age. Several studies have demonstrated that the overall risk of sudden death in asymptomatic patients with aortic stenosis is around 2%. Once symptoms develop, there is an inexorable deterioration with a poor prognosis. Within 3 years of the onset of angina, syncope, or the symptoms of heart failure, 75% of symptomatic patients are dead unless the outflow obstruction is relieved. Therefore, the modality to solve AS is life saving for this patient group. Before 2002 when first-in-man transcatheter aortic valve implantation (TAVI) was performed, surgical aortic valve replacement (SAVR) is the only treatment of choice for patients with severe symptomatic aortic stenosis. As TAVI prevailed, TAVI has been demonstrated to be safe and effective in relieving AS in patients with high and intermediate surgical risk. Transfemoral approach is preferential approach of TAVI. As the device evolved, transfemoral TAVI procedure is moving to local anaesthetic with percutaneous procedure instead of surgical cut-down.

Femoral arteriotomy closure following TAVI remains challenging and, at times, may result in significant or even fatal complications. Even though the evolution of device and smaller device size, complications associated with the femoral access site are reported in 5-20% of patients undergoing TAVI. The incidence of access site-related vascular complications reinforces the need for the improvement of techniques that ensure effective and reproducible hemostasis with a safe and effective arteriotomy closure. The Perclose ProGlide (PP) suture-mediated closure device (Abbott Vascular, Santa Clara, CA, USA) has been widely utilized in a dual pre-close strategy, and successful closures may be obtained for up to 24F sheath. Moreover, the preclose technique has been shown not to increase the risk of CFA narrowing. Therefore, the preclose technique has been widely used in percutaneous endovascular procedures using large diameter arteriotomies, including TAVI and EVAR.

Nevertheless, failure of this device requiring further intervention has been described in 4-9% of cases. Adjunctive Angio-Seal technique has been postulated as feasible and safe or even considered as a bail-out strategy when the dual PP closure technique fails to obtain complete hemostasis. Therefore, the best strategy for femoral arteriotomy closure following TAVI remains to be studied.

In our hospital, we have performed either dual PP or one Perclose ProGlide with one Angio-Seal for femoral arteriotomy closure following TAVI. Both have been shown to be satisfactory for complete hemostasis. However, there was not study regarding complete hemostasis, long-term vessel outcome and clinical walking ability between these two procedures. Herein, we design a open-labeled randomized study to compare the efficacy of complete hemostasis and long-term vascular outcome between dual PP and one Perclose ProGlide with one Angio-Seal following TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 20 years old
* Severe aortic stenosis and suitable candidate for transfemoral transcatheter aortic valve implantation

Exclusion Criteria:

* Age < 20 years old
* Severe aortic stenosis not suitable for transfemoral transcatheter aortic valve implantation
* An initial plan for a surgical transfemoral cut-down approach

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Vascular complication | during hospitalization for index procedure
  TAVI related major or minor vascular complication according to valve academic research consortium 3 criteria
Life threatening bleeding complication | within 24hrs after the index procedure
  TAVI related life threatening bleeding according valve academic research consortium 3 criteria
Major or minor bleeding complication without life threatening condition | within 24hrs after the index procedure
  TAVI related major or minor bleeding according valve academic research consortium 3 without life threatening condition

SECONDARY OUTCOMES:
Bail-out closure device use | within 10mins after the index procedure
  additional closure device deployment for femoral access site to achieve hemostasis
Limb ischemia related to TAVI | within one year after TAVI
  Significant peripheral ischemia related to arteriotomy closure
In-hospital serious vascular complications requiring percutaneous or surgical interventions | In the index hospitalization (up to 14 days)
  Vascular perforation or dissection, peripheral ischemia or acute limb ischemia, arteriovenous fistula, pseudoaneurysm, and access-site hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Mao-Shin Lin, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yeh CF, Kao HL, Ko TY, Chen CK, Tsai CH, Huang CC, Chen YH, Chan CY, Lin MS. Dual ProGlide vs ProGlide and Angio-Seal for Femoral Access Hemostasis After Transcatheter Aortic Valve Replacement: A Randomised Comparative Trial. Can J Cardiol. 2025 Jan;41(1):12-20. doi: 10.1016/j.cjca.2024.09.001. Epub 2024 Sep 6. PMID 39245341